CLINICAL TRIAL: NCT01277848
Title: PLAC1 in Reproduction
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: March of Dimes (Other)
Responsible Party: Principal Investigator, Michael Fant, Principal Investigator, University of South Florida
Other Study IDs: IRB#107849
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Pregnancy
Keywords: PLAC1; pregnant; first prenatal visit; pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The PLAC1 gene is a recently described X-linked gene that maps to a region of the X chromosome thought to be important for normal fetal and placental development. Elevated levels of PLAC1 mRNA were detected in preeclampsia and appeared to be directly related to disease severity. PLAC1 may serve as a useful marker of placental dysfunction or threatened pregnancy.

The objective of this study is to measure the prevalence of circulating anti-PLAC1 antibodies in pregnant maternal serum and correlate it with pregnancy outcome. It is likely that women with these antibodies are at higher risk for adverse pregnancy outcomes. Approximately 5% (50 of 1000) will be expected to have anti-PLAC1 antibodies based on previously reported data. The prevalence of these antibodies and their clinical impact on pregnancy outcomes will be determined.

1000 healthy, multiparous and primigravid women will be screened for anti-PLAC1 antibodies at their routine prenatal clinic visits. Subjects will be enrolled at their first clinic visit at USF Health, South Tampa Center, Department of Obstetrics. Blood (1.0 ml) will be obtained as part of the routine blood draw at the time of enrollment. Blood will only be collected when drawn as part of routine laboratory testing as determined by the primary care provider.

Additional blood samples (1.0 ml) will be collected throughout pregnancy at the same time blood is obtained for routine or otherwise clinically indicated laboratory testing. A maximum of 5 samples will be collected through the pregnancy.

Maternal demographic data will be collected and patients will be followed longitudinally to the completion of pregnancy to ascertain their clinical status during pregnancy, onset of premature labor, premature rupture of membranes, delivery date, and gestational age at delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, primigravid and multigravid women between the ages of 14 and 55, receiving prenatal care at USF Health, STC, Dept. of Obstetrics.

Exclusion Criteria:

* presence of significant cardiac disease
* renal disease
* chronic hypertension
* chromosomal abnormalities
* cancer

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women at USF coming in for their first prenatal appointment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2009-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Anti-PLAC1 autoantibodies | During pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fant, MD, PhD, Principal Investigator — University of South Florida
Locations (1):
- USF Health OB/GYN Clinic, Tampa, Florida, United States